CLINICAL TRIAL: NCT03156868
Title: Analysis of Soluble Mediators, Cytokines, and Circulating Angiogenic Factors (FACs) as Potential Predictors / Prognostic Factors in Antiangiogenic Therapy Following Failure of First-line Chemotherapy in Advanced Non-squamous Lung Carcinoma
Brief Title: Analysis of Soluble Mediators,Cytokines and FACs as Prognostic Factors in Advanced Non-squamous Lung Carcinoma
Status: Completed | Type: Observational
Sponsor: Spanish Lung Cancer Group (Other)
Responsible Party: Sponsor
Other Study IDs: GECP 16/02_SELINA
Record Dates: First submitted 2017-05-12; First posted 2017-05-17 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Soluble mediators analyzed (cytokines, FACs)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Recent studies have shown that the assessment of a set of cytokines and / or circulating angiogenic factors (FACs) could be used to identify prognostic factors predictive of efficacy and / or potential mechanisms of resistance to antiangiogenic agents

DETAILED DESCRIPTION:
Current management of patients with locally advanced or metastatic NSCLC, with no susceptible molecular alterations (EGFR mutation, ALK translocation, ROS1 fusion), includes combinations based on platinum in the first line of treatment, while in the second Line, there are three possibilities in monotherapy: docetaxel, erlotinib and pemetrexed. Pemetrexed is exclusively indicated for patients with a NSCLC of non-squamous histology. Although all of them have been shown to increase progression-free survival (PFS) and overall survival (OS), the median time to progression is maintained at 3 months, and the median overall survival at 8-9 months.

Recently, other therapeutic options have been incorporated in the context of the second line. Firstly, two antiangiogenic drugs: nintedanib and ramucirumab. The combination of nintedanib or ramucirumab with docetaxel in the second line of treatment has been shown to provide a significant increase in SLP and SG compared to docetaxel (9,11). One of the criticisms of the results of these two trials, common to all antiangiogenic treatments, is the lack of predictive factors that help us to better select the patients who would benefit from such treatment, as well as a better rationalization of Economic costs. On the other hand, recent data from new strategies based on immunotherapies in lung cancer indicate that nivolumab, a PD-1 antibody (Programmed cell death-1), has shown benefit in terms of survival versus docetaxel monotherapy both in Histology as squamous adenocarcinoma after failure to a platinum-based prior line.

Based on the above, the objective of this project is to analyze a panel of soluble mediators by means of multiparametric immunoassay techniques in samples of peripheral blood (at baseline, during treatment, and progression of the disease) obtained from patients With advanced lung adenocarcinoma, without molecular alterations treatable with anti-target drugs, that have progressed to a first line of chemotherapy, irrespective of whether they have received treatment with immunotherapies, and that they will be treated in the second line with chemotherapy (docetaxel) In combination or not with an antiangiogenic. It is a question of analyzing markers or panels of them with a prognostic / predictive meaning, as well as those that could be related to mechanisms of resistance to the administered treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 years
2. Histological and / or cytological confirmation of non-squamous pulmonary carcinoma, stage IIIB / IV or recurrent
3. Failure to a first line of chemotherapy for advanced or recurrent disease. Patients who have received 2 treatment lines will also be included and this will be the 3 rd line provided that during one of the previous lines they have received immunotherapy or antidandial therapies (in patients with a wild type or unknown mutational status).
4. ECOG 0 or 1
5. Life expectancy greater than 12 weeks.
6. Written informed consent of the patient in accordance with current regulations

Exclusion Criteria:

1. Receive more than one line of chemotherapy treatment for advanced disease
2. Hepatic function (one or more of the following values would exclude the patient): a. Total bilirubin outside the limits of normality; B. For patients without hepatic metastasis: ALT or AST> 1.5 times ULN; C. For patients with hepatic metastases: total bilirubin outside the limits of normality, ALT or AST> 2.5 times the ULN.
3. Hemogram (one or more of the following values would exclude the patient): a. Absolute neutrophil count <1,500 / mm3; B. Platelets <100,000 / mm 3; C. Hemoglobin <9.0 g / dl.
4. Situations such as the following: a. Active serious infections, especially if they require antimicrobial or systemic antibiotic treatment, or active or chronic infection with hepatitis C or B virus; B. Severe disease or non-oncological concomitant disease such as neurological, psychiatric or infectious disease or active ulcers (digestive tract, skin) or relevant analytical abnormality; C. Patients who are sexually active and do not want to use a medically acceptable method of contraception during the study and for at least 3 months after the completion of active treatment; D. Psychological, family, sociological or geographical factors; and. Alcoholism or current drug addiction; F. Preexisting ascites and / or clinically significant pleural effusion; G. Decompensated diabetes mellitus or other contraindication to treatment with corticosteroids at high doses
5. Pregnancy or breastfeeding; The women must have obtained a negative result in a pregnancy test before starting the treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced non-squamous lung carcinoma without molecular alterations susceptible to be treated with specific inhibitors (EGFR mutation, ALK translocation, ROS1 fusion) that have progressed to the first line of chemotherapy and are subsidiary to a second treatment line.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2016-08-03 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Soluble mediators in relation to progression free survival | At time of progression, an average of 1 year
  to correlate soluble mediators at progression time

SECONDARY OUTCOMES:
Soluble mediators in relation to response rate | at time of first response, an average of 3 months
  the soluble mediators will be measured in the blood sample at time of first response

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Camps, MD, Principal Investigator — Hospital General Universitario de Valencia
Locations (25):
- Spain (25):
  - Hospital de Elche, Elche, Alicante
  - Hospital de Torrevieja, Torrevieja, Alicante
  - ICO-Badalona, Badalona, Barcelona
  - Hospital General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Complejo Hospitalario Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria, Gran Canaria
  - Hospital Severo Ochoa, Leganés, Madrid
  - Hospital Son Llàtzer, Palma de Mallorca, Mallorca
  - Hospital Costa del Sol, Marbella, Málaga
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Universitario de la Ribera, Alzira, Valencia
  - H.G.U. Alicante, Alicante
  - Hospital Universitari Quirón Dexeus, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - H. Provincial de Castellón, Castelló
  - Hospital de Jaén, Jaén
  - Hospital Lucus Agustí, Lugo
  - H.U. Puerta de Hierro, Madrid
  - H. Clínico San Carlos, Madrid
  - Hospital Clinico de Salamanca, Salamanca
  - Hospital Nuestra Señora Candelaria, Santa Cruz de Tenerife
  - Hospital Sant Pau i Santa Tecla, Tarragona
  - H. General U. de Valencia, Valencia
  - Hospital Dr. Peset, Valencia
  - Hospital de Sagunto, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org